CLINICAL TRIAL: NCT06853600
Title: Optimización Del Rendimiento Durante El Entrenamiento De Fuerza a Través De Implementación Aguda De Suplementación Nutricional
Brief Title: Effects of Rhodiola Rosea Supplementation on Mental Fatigue, Visuo-cognitive Processing, and Strength Performance
Acronym: Rhodiola Rosea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Amador García Ramos, Head of Research Group, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SICEIA-2024-000283
Record Dates: First submitted 2025-02-20; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Sport Medicine
Keywords: Adaptogens; Fatigue; Sports supplementation; Strength training; Rhodiola Rosea; Visuo-cognitive Processing; Triple-Blinded Randomized Placebo Crossover Study
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rhodiola Rosea and mental fatigue (Experimental)
  Interventions: Dietary Supplement: Rhodiola Rosea Capsules
- Rhodiola Rosea and no fatigue (Experimental)
  Interventions: Dietary Supplement: Rhodiola Rosea Capsules
- Placebo and mental fatigue (Experimental)
  Interventions: Dietary Supplement: Rhodiola Rosea Capsules
- Placebo and no fatigue (Experimental)
  Interventions: Dietary Supplement: Rhodiola Rosea Capsules

INTERVENTIONS:
Dietary Supplement: Rhodiola Rosea Capsules — One of the most practical and accessible options for mitigating the occurrence of mental fatigue is the strategic use of nutritional supplements. Several nutritional supplements have been shown to reduce behavioural or subjective markers of mental fatigue, including caffeine, creatine, panax ginseng, and various vitamins or minerals. Among these, Rhodiola Rosea (RR), a supplement with purported adaptogenic and ergogenic properties, has gained attention. Several randomized controlled trials have reported reductions in mental fatigue after RR supplementation without adverse effects. The main objective of this study was to explore the effects of four days of Golden Root Extract (RR) supplementation on mental fatigue, visuo-cognitive processing, strength performance, and perceived exertion in young, healthy individuals.

SUMMARY:
This document aims to provide information to request authorization to collect data on the effects of supplementation administered 30 minutes before resistance training on the number of repetitions, execution speed, and perceived effort for the bench press and bench pull exercises. To grant authorization, an informed consent form must be signed for the use of the information.

If authorization is granted, personalized information will be provided by the professional requesting the consent. It is recommended to read this document beforehand and ask any questions necessary to understand the details. If desired, the document can be taken for consultation with others, allowing ample time to make a decision.

The decision is entirely voluntary. It is possible to decline authorization for the use of personal and/or health data without affecting the relationship with the professional requesting the consent or healthcare services.

PURPOSE OF THIS REQUEST Participation involves attending a total of 5 sessions. The study begins with a familiarization session, which includes measurements of weight, height, and the determination of the 20-repetition maximum load (i.e., the maximum load that can be lifted between 18-22 times), which will be used in the rest of the experimental sessions. In the experimental sessions, a supplement capsule will be administered 30 minutes before starting the resistance training. The composition of the capsule will not be disclosed to ensure a triple-blind approach for participants and evaluators.

The resistance training will consist of 4 supersets (each superset consisting of two exercises: bench press and bench pull). There will be 5-minute breaks between each superset and 1.5-minute breaks between the two exercises within the same superset. During the supersets, the maximum number of repetitions will be performed until reaching muscle failure. Heart rate and blood pressure will be measured during the training, and perceived effort will be recorded. No physiological samples will be collected. This study aims to provide a clearer understanding of which supplement may have the most beneficial effects when training with light loads and repetitions to failure in a superset, a topic that has not been explored before.

REQUEST DETAILS The professional attending to this study is Amador García Ramos. By signing this document, authorization is given to complete questionnaires about perceived effort.

POTENTIAL BENEFITS AND RISKS No specific benefits or risks are expected. Participation will contribute to increasing scientific knowledge.

No compensation will be provided for authorizing the use of health data. Additionally, the researchers involved in this project will not receive specific compensation for their participation in the study.

DETAILED DESCRIPTION:
The current study is a randomized, placebo-controlled, triple-blind (participants, researchers, and data analysts), and crossover experimental trial. Participants visit the laboratory on five occasions separated by seven days: one preliminary testing session and four experimental sessions. During the preliminary testing session, participants are introduced to the Stroop and MOT tests, followed by the determination of 1RM loads for the bench press and bench pull exercises.

The four experimental sessions follow the same protocol, differing only in the supplement (Rhodiola Rosea [RR] or placebo) and mental task conditions (Stroop test or control video). Participants are counterbalanced and assigned to each experimental session condition using the Research Randomizer online software (www.randomizer.org): (I) RR and Stroop test, (II) RR and control video, (III) placebo and Stroop test, and (IV) placebo and control video.

The assessment order in each experimental session is as follows: (I) mental task condition (Stroop test or control video), (II) MOT pre-training, (III) strength training, and (IV) MOT post-training. All sessions are conducted on the same day of the week and at consistent times (±1 hour) for each participant. Participants are instructed to avoid stimulants on the testing day and refrain from resistance exercise 24 hours before the visit.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* At least one year of resistance training experience
* Ability to execute the bench press and bench pull exercises at maximal intentional velocity with proper technique

Exclusion Criteria:

- Any medical condition that could impede proper engagement in resistance training

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-05-25 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Strength training | During training
  The general warm-up mirrored that of the 1RM assessment. Thereafter, the specific warm-up included for each exercise 2 sets of 3 repetitions at 30% and 50% of 1RM, and a final set of 2 repetitions at 70% of 1RM. The training regimen consisted of 8 alternating sets (4 sets each) of bench press and bench pull, with a 2-minute rest period between sets, performed at 70% of the 1RM load established during the preliminary testing session. Sets were terminated when 2 consecutive repetitions were performed at a MV below 0.35 m·s-1 for the bench press and 0.60 m·s-1 for the bench pull. Participants were encouraged to perform all repetitions at maximal intent, and they received real-time MV feedback (GymAware RS; Kinetic Performance Technologies, Canberra, Australia). Strength performance was assessed by recording the number of repetitions completed (Nrep) and the velocity of the fastest repetition (MVfastest) in each set.
  The OMNI-Resistance Exercise Scale (OMNI-RES) of perceived exertion was

SECONDARY OUTCOMES:
MOT test | Baseline (before training) and immediately after training
  In line with the method used by Vera et al. [26] for the MOT test, eight identical black balls (each with a diameter of 1.8 cm) were displayed on a white square background (32.5 cm, luminance of 107 cd/m²) subtending a visual angle of 36°. The stimuli were presented on a 27-inch television monitor (LS27C330GAUXEN) positioned 50 cm away from the participant. At the beginning of each trial, three of the balls were randomly illuminated in green for 2 seconds, after which they reverted to their original black colour. Participants were instructed to track the selected balls for a duration of 10 seconds. No specific strategy was suggested for completing the task, and participants were allowed to use natural eye movements, mirroring real-world scenarios [27,28]. None of the participants had prior experience with the MOT task. The balls moved along linear paths at a constant speed, changing direction only when colliding with each other or the walls.
  After the 10-second tracking period, all t
Cognitively demanding and control tasks | Baseline (before training)
  A 30-minutes incongruent Stroop task was used to induce mental fatigue, which requires response inhibition and sustained attention [24] and has demonstrated to be a valid intervention for inducing mental fatigue and impairing physical performance [1,25]. In the incongruent Stroop colour word task, participants were shown lists of colour words (e.g., "blue", "red", "yellow", or "green") on the screen, where the ink colour of the letters did not match the word itself (for example, the word "blue" might be displayed in green ink). For each word, participants were instructed to select the ink colour rather than reading the word. After each response, a new word was presented. The control condition consisted of watching an emotionally neutral documentary during 30 minutes in the same screen (LS27C330GAUXEN, 27", Samsung, Seoul, Korea) used for the Stroop task. Participants remained seated in the same room and in the same position for both interventions (50 cm from the screen).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport Science, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shevtsov VA, Zholus BI, Shervarly VI, Vol'skij VB, Korovin YP, Khristich MP, Roslyakova NA, Wikman G. A randomized trial of two different doses of a SHR-5 Rhodiola rosea extract versus placebo and control of capacity for mental work. Phytomedicine. 2003 Mar;10(2-3):95-105. doi: 10.1078/094471103321659780. PMID 12725561
- [Background] Spasov AA, Wikman GK, Mandrikov VB, Mironova IA, Neumoin VV. A double-blind, placebo-controlled pilot study of the stimulating and adaptogenic effect of Rhodiola rosea SHR-5 extract on the fatigue of students caused by stress during an examination period with a repeated low-dose regimen. Phytomedicine. 2000 Apr;7(2):85-9. doi: 10.1016/S0944-7113(00)80078-1. PMID 10839209
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12725561/